CLINICAL TRIAL: NCT06055816
Title: Gemcitabine Combined With Endostar and Envafolimab in Elderly Patients With Locally Advanced Nasopharyngeal Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Chen Xiaozhong, Professor, Zhejiang Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GEE study
Record Dates: First submitted 2023-08-14; First posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — endostar protein; envafolimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gemcitabine Combined With Endostar and Envafolimab (Experimental): Neoadjuvant therapy consisting of gemcitabine (1000mg/m2 d1,8) , endostar (150mg 3-day continuous infusion) and envafolimab (240mg d1) was given every 3 weeks for 3 cycles. Endostar, administered every 3 weeks (150mg 3-day continuous infusion), was given concurrently with intensity-modulated radiotherapy.
  Interventions: Drug: Endostar and Envafolimab

INTERVENTIONS:
Drug: Endostar and Envafolimab — Neoadjuvant therapy consisting of gemcitabine (1000mg/m2 d1,8) , endostar (150mg 3-day continuous infusion) and envafolimab (240mg d1) was given every 3 weeks for 3 cycles. Endostar, administered every 3 weeks (150mg 3-day continuous infusion), was given concurrently with intensity-modulated radiotherapy.

SUMMARY:
Gemcitabine Combined With Endostar and Envafolimab in Elderly Patients With Locally Advanced Nasopharyngeal Carcinoma

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥65 years with newly pathologically confirmed NPC
* Karnofsky performance status ≥60
* Clinical stage III-IVA (Union for International Cancer Control and American Joint Committee on Cancer staging system for NPC, 8th edition)
* Adequate organ function

Exclusion Criteria:

* Cancer history
* Prior radiotherapy, cytotoxic chemotherapy, immunotherapy or target therapy
* Life-expectance within 6 months

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-09-28 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients with grade 3 or higher adverse events (AEs). | Up to 24 weeks
  The primary endpoint was the safety profile. AEs were scored according to the Common Terminology Criteria for Adverse Events (CTCAE) v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Xiaozhong Chen, Principal Investigator — Department of Radiation Oncology, Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided